CLINICAL TRIAL: NCT06721312
Title: Continuous Heart Rate Variability Monitoring in Doctors; Understanding Patterns of Stress and Recovery and Their Relationship With Self-reported Resilience, Burnout and Wellbeing.
Acronym: HEART-ED
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-015-24
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Burnout; Burnout Syndrome; Occupational Stress; Stress
Keywords: Heart rate variability; HRV; occupational stress; resilience; fatigue; wellbeing; stress; burnout
MeSH Terms: conditions — Burnout, Psychological; Occupational Stress; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Burnout is an increasing concern in the medical professions. This study aims to utilise established, validated self-report measures combined with continuous heart rate variability measurements to better understand the stress and recovery patterns experienced by doctors that may contribute to burnout.

This mixed methods study design will consist of an ecological momentary assessment phase where participants will complete commonly used and validated real-time subjective measures while concurrently wearing a heart rate variability monitor to provide an objective measure of stress. Following on from this, participants of interest will be invited to participate in semi structured interviews to further explore their experiences of stress and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Working within NHS Grampian
* Access to a smartphone

Exclusion Criteria:

* Cardiac arrhythmias/endocrine disease.
* Prescription beta blockers, calcium channel blockers, ACE inhibitors, benzodiazepines, antidepressants and antianxiety medications.
* Insufficient non-working time prior to study commencement.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical Doctors working within NHS Grampian
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 7 days
  Continuous heart rate variability over 7 day study period

SECONDARY OUTCOMES:
Burnout | Measured on day 1
  Maslach Burnout Inventory -
  22 item scale measuring occupational burnout. Each item asks participants to rank on a scale from never to every day. An overall score is then calculated from the results.
Resilience | Measured on day 1
  Resilience Scale for Adults The RSA is a 33-item self-report scale examining intrapersonal and interpersonal factors presumed to assist them to be able to adapt to adversities. Responses are provided via 5-point Likert scale.
Wellbeing | Measured on day 1
  ICOPPE Wellbeing Scale The I-COPPE scale(21) has 6 individual domains of interpersonal, community, occupational, physical, psychological, and economic - all of which have been individually validated against overall wellbeing. The scale asks participants to rate each of the wellbeing domains at three different time points, now, one year previously and one year in the future totalling 21 items.
EMA Measures | 8 times/day for 7 days
  Real-Time Job Demands NASA task load index (NASA TLX) is a multidimensional workload assessment tool. It contains six subscales of mental demand, physical demand, temporal demand, performance, effort, and frustration. The overall workload is derived from an average of the six subscales listed.
  Real-Time Job Resources This is a six-item scale derived from the job-demands resources model of burnout. The items contained within the scale are feedback, rewards, job control, participation, job security and supervisor support.
  Flow Included is a single item question asking participants "have you felt completely absorbed by a challenging but doable task". Given the paucity of literature understanding what "flow" might mean within this study population and how this may relate to HRV there is a free text box allowing participants to expand on their experience.
  Fatigue The Rating of Fatigue (ROF) scale(59)is a single-item visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Grampian, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kane L, Ball D, Martin KR, Powell D. Continuous heart rate variability monitoring-understanding patterns of stress and recovery and their relationship with self-reported burnout, resilience and well-being in doctors: a protocol for a sequential explanatory mixed-methods study. BMJ Open. 2025 Jun 8;15(6):e097849. doi: 10.1136/bmjopen-2024-097849. PMID 40484420